CLINICAL TRIAL: NCT05379907
Title: Observational Study of ctDNA in Resectable and Borderline Resectable Pancreatic Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Determined that the tumor analysis could not be performed in accordance with the protocol.
Sponsor: Inova Health Care Services (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: U22-02-4671
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients who have been diagnosed with R/BR PDAC and who have residual formalin-fixed paraffin-embedded (FFPE) tissue available will provide FFPE and whole-blood samples for SIGNATERA™ testing at baseline. Patients will provide additional whole-blood samples for SIGNATERA™ testing at months 1, 2, 4, 6, 9, 12, and 15 from the date of informed consent. The blood samples will be stored at the Inova Schar Cancer Institute and may be shared for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SIGNATERA™ ctDNA testing — Information collection about how SIGNATERA™ ctDNA testing changes how doctors make treatment recommendations to patients with early-stage pancreatic cancer.

SUMMARY:
The purpose of this study is to collect information about treatment recommendations based on ctDNA testing and whether treatment changes based on ctDNA information result in better outcomes for patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Resectable or borderline resectable pancreatic adenocarcinoma per NCNN guidelines
3. No prior radiation therapy, chemotherapy, targeted therapy, investigational therapy, or surgery for pancreatic cancer.
4. ECOG performance status ≤ 1
5. Clinically eligible for chemotherapy
6. Able to tolerate collection of up to 20 mL of blood via venipuncture for research blood draw
7. Has residual FFPE specimen available for submission to Natera
8. Able to read, understand and provide written informed consent
9. Willing and able to comply with the study requirements

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Radiologic evidence of distant metastases
3. Prior history and treatment for any cancer within the past year or has another active cancer, with the exception of non-melanoma skin cancer
4. Prior initiation of chemotherapy, radiation therapy, or surgery for pancreatic cancer
5. Neuropathy > grade 2
6. History of bone marrow or organ transplant
7. Blood transfusion within 1 month of enrollment
8. Medical condition that would place the patient at risk as a result of blood donation, such as bleeding disorder
9. Serious medical condition that may adversely affect ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants with Resectable and Borderline Resectable Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Impact of SIGNATERA™ on treatment decisions | 2 years
  Examine the impact of SIGNATERA™ on treatment decisions as determined by physician questionnaires

SECONDARY OUTCOMES:
Frequency of positive SIGNATERA™ ctDNA testing | 2 years
  Determine the frequency of positive SIGNATERA™ ctDNA testing in patients with R/BR PDAC at baseline and after surgical resection
Overall survival of patients managed with SIGNATERA™ ctDNA data | 2 years
  Compare overall survival of patients managed with available SIGNATERA™ ctDNA data to historical controls
Progression-free survival of patients managed with SIGNATERA™ ctDNA data | 2 years
  Compare progression-free survival of patients managed with available SIGNATERA™ ctDNA data to historical controls
Patient satisfaction of SIGNATERA™ ctDNA on treatment recommendations | 2 years
  Assess patient satisfaction regarding the potential role of SIGNATERA™ ctDNA on treatment recommendations using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Wadlow, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Pancreatic Cancer Collaborators. The global, regional, and national burden of pancreatic cancer and its attributable risk factors in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2019 Dec;4(12):934-947. doi: 10.1016/S2468-1253(19)30347-4. Epub 2019 Oct 21. PMID 31648972
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Varadhachary GR, Tamm EP, Abbruzzese JL, Xiong HQ, Crane CH, Wang H, Lee JE, Pisters PW, Evans DB, Wolff RA. Borderline resectable pancreatic cancer: definitions, management, and role of preoperative therapy. Ann Surg Oncol. 2006 Aug;13(8):1035-46. doi: 10.1245/ASO.2006.08.011. Epub 2006 Jul 24. PMID 16865597
- [Background] Spitz FR, Abbruzzese JL, Lee JE, Pisters PW, Lowy AM, Fenoglio CJ, Cleary KR, Janjan NA, Goswitz MS, Rich TA, Evans DB. Preoperative and postoperative chemoradiation strategies in patients treated with pancreaticoduodenectomy for adenocarcinoma of the pancreas. J Clin Oncol. 1997 Mar;15(3):928-37. doi: 10.1200/JCO.1997.15.3.928. PMID 9060530
- [Background] Philip PA, Lacy J, Portales F, Sobrero A, Pazo-Cid R, Manzano Mozo JL, Kim EJ, Dowden S, Zakari A, Borg C, Terrebonne E, Rivera F, Sastre J, Bathini V, Lopez-Trabada D, Asselah J, Saif MW, Shiansong Li J, Ong TJ, Nydam T, Hammel P. Nab-paclitaxel plus gemcitabine in patients with locally advanced pancreatic cancer (LAPACT): a multicentre, open-label phase 2 study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):285-294. doi: 10.1016/S2468-1253(19)30327-9. Epub 2020 Jan 14. PMID 31953079
- [Result] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Result] Dasari A, Morris VK, Allegra CJ, Atreya C, Benson AB 3rd, Boland P, Chung K, Copur MS, Corcoran RB, Deming DA, Dwyer A, Diehn M, Eng C, George TJ, Gollub MJ, Goodwin RA, Hamilton SR, Hechtman JF, Hochster H, Hong TS, Innocenti F, Iqbal A, Jacobs SA, Kennecke HF, Lee JJ, Lieu CH, Lenz HJ, Lindwasser OW, Montagut C, Odisio B, Ou FS, Porter L, Raghav K, Schrag D, Scott AJ, Shi Q, Strickler JH, Venook A, Yaeger R, Yothers G, You YN, Zell JA, Kopetz S. ctDNA applications and integration in colorectal cancer: an NCI Colon and Rectal-Anal Task Forces whitepaper. Nat Rev Clin Oncol. 2020 Dec;17(12):757-770. doi: 10.1038/s41571-020-0392-0. Epub 2020 Jul 6. PMID 32632268